CLINICAL TRIAL: NCT06323876
Title: The Role of Quantitative CT and Radiomic Biomarkers for Precision Medicine in Pulmonary Fibrosis
Acronym: Radiomics
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Imre Noth, MD, Department Chair of Pulmonary & Critical Care, University of Virginia
Other Study IDs: HSR231590; R01HL171918 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: CT; biomarkers; gene expression; radiomic markers
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens are blood DNA, RNA, and plasma proteins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- University of Chicago: This cohort will have prior consent to the Natural History of Interstitial Lung Disease, which is an ongoing, longitudinal cohort of patients with clinically diagnosed ILD, including IPF. Patients are recruited from University of Chicago Interstitial Lung Disease Program during their clinic visit. Blood, plasma, and serum samples are collected upon enrollment and stored in a biorepository at University of Chicago. Subsets of patients have repeat blood draw at return clinic visits for specific research studies. The investigators propose collection of 1-year HRCTs, FVC, and DLCO.
  Interventions: Diagnostic Test: HRCT; Diagnostic Test: Blood Draw
- University of Virginia: This cohort will have prior consent to the Natural History of Interstitial Lung Disease, which is an ongoing, longitudinal cohort of patients with clinically diagnosed ILD, including IPF. Patients are recruited from the UVA Interstitial Lung Disease Program during their clinic visit. Blood, plasma, and serum samples are collected upon enrollment and stored in a biorepository at UVA (Pinn Hall RM#2232B, IRB#20937). Subsets of patients have repeat blood draw at return clinic visits for specific research studies. The investigators propose collection of 1-year HRCTs, FVC, and DLCO.
  Interventions: Diagnostic Test: HRCT; Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: HRCT — High resolution computed tomography (HRCT) scan is a medical imaging technique used to obtain detailed internal images of the body. HRCT images will be obtained at 0 and 12 months.
Diagnostic Test: Blood Draw — During blood draw, someone uses a needle to take blood from a vein, usually in your arm.

SUMMARY:
This observational study involves obtaining 2 chest CT scans; a historical baseline CT within ±1 year of enrollment into PRECISIONS, and a follow-up CT (either historical or prospective) 12 months ± 180 days after the baseline CT. Many IPF patients will have a CT scan every 12 months for disease monitoring and cancer screening. Participants will have the option to share historical CTs only or they can choose to have a research CT done for the follow-up scan, if a scan for clinical purposes is not available.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) remains deadly despite two FDA-approved therapies. Forced vital capacity (FVC), a one-dimensional assessment of lung function that requires three effort-dependent and error-prone maneuvers, is the standard for evaluating disease severity and monitoring progression. FVC indirectly measures disease activity and is thus insensitive to subtle change. These limitations hamper therapeutic trials. The Gender, Age, and Physiology (GAP) score improves on FVC alone and is the most used scoring model for prognostication, but gender and age aren't influenced by treatment. Modifiable intermediate molecular markers and other metrics for assessing disease severity and progression remain unmet needs for aiding drug development and clinical decision-making. Computed tomography (CT) captures morphologic patterns and the extent of fibrosis noninvasively. Advances in quantitative CT enable objective detection and quantitation of anatomy, and highly dimensional image features, often termed radiomic, can identify sub-visual characteristics. The investigators seek to evaluate radiomic features alone and in conjunction with other disease dimensions for prognostication and response to treatment in IPF.

The investigators overall objectives are to identify and validate radiologic features, such as total extent of lung fibrosis, for disease activity and intermediate response to therapy, and understand where to position these powerful markers. The investigators hypothesize that DTA scores will contribute to prediction of disease progression and that molecular markers will enhance that performance.

Aim 1: The investigators will validate quantitative CT and radiomic markers for disease progression by independent replication in separate cohorts. The investigators hypothesize that quantitative CT markers will predict disease progression in UVA/Chicago cohorts. Baseline and subsequent CT scans have been voluntarily collected in many PFF-PR cases. The investigators propose collection of 1-year HRCTs in UVA/Chicago participants to evaluate: a) the prognostic value of baseline quantitative CT and radiomic markers (i.e. DTA) in predicting time to progression defined as either 10% relative decline in FVC, lung transplant, or death from any cause, b) associations between changes in CT biomarkers on sequential CT and changes in 1-year FVC and DLCO, and c) change in CT associated with drug treatment. This aim will establish the relative and synergistic value of CT to established physiologic markers.

Aim 2: The investigators will determine if candidate genetic variants for IPF susceptibility and survival are associated with the DTA score and improve predictive performance for survival. The investigators hypothesize that variants in MUC5B, TOLLIP, and Telomere lengths (TL) will enhance DTA fibrosis score associations with progression-free survival in IPF. The investigators will perform a cross-sectional analysis of PFF-PR cases comparing quantitative CT and radiomic markers at baseline with and without "at risk" genotypes for association with severity and progression (decline in FVC over time). This will ascertain what markers improve performance of the DTA fibrosis extent scores using Cox regression analysis and accuracy metrics from Aim 1. Findings will be replicated in UVA/Chicago cohort and in the prospective PRECISIONS cohort. This aim will establish the additive value of genetic markers.

Aim 3: The investigators will assess whether DTA and radiomic markers are additive/synergistic with plasma protein and blood transcriptome markers for disease progression. The investigators hypothesize that selected protein and transcriptomic markers will prove additive to DTA fibrosis extent for prediction of progression-free survival whereas other markers correlated with DTA will not. The investigators have chosen published markers from a 4-protein panel signature, along with CCL18, as examples, given their current level of replication and promise. The investigators will also include a 25-gene FVC predictor for disease progression. Similar analyses, as outlined in Aims 1 and 2, will determine their additive information value.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 40 years of age
2. Diagnosed with IPF according to 2018 ATS/ERS/JRS/ALAT confirmed by the enrolling investigator
3. Signed informed consent

Exclusion Criteria:

1. Pregnancy or planning to become pregnant
2. Women of childbearing potential not willing to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year during study participation*
3. Significant medical, surgical or psychiatric illness that in the opinion of the investigator would affect subject safety or potential to complete the research study

   * A woman is considered to be of childbearing potential if she is post-monarchical, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

Ages: 40 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Pulmonary Fibrosis as described above in inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Derivation of DTA in IPF only cases from the PFF-PR and its associations with disease severity and outcomes. | 12 months
  Driven texture analysis (DTA) is a machine learning method capable of automatic detection and quantification of lung fibrosis on HRCT. It is trained to discriminate fibrosis using radiologist-identified image regions demonstrating normal lung parenchyma and usual interstitial pneumonia patterns.
  Changes in Forced Vital Capacity (FVC) measured in liters, reflect increased elastic recoil caused by fibrosis. We will use linear-mixed effects models with random intercept to examine associations of repeated DTA-fibrosis scores with repeated percent predicted FVC measurements over time (12 months minimum). This approach will provide a more precise estimate, power, and account for baseline FVC at an individual level which has implications of how rapid a decline we anticipate. This is the most common approach to examine longitudinal changes of FVC in IPF studies. FVC decline greater than 10% has been shown to be prognostic of worse survival and is a common endpoint in IPF clinical trials.
Determine whether known IPF-risk genetic variants are associated with DTA score. | 12 months
  This is a cross-sectional analysis to determine whether genetic variants that confer higher risk of disease and progression are associated with higher DTA scores from CT.
Identify novel genetic variants that associate with DTA score progression. | 12 months
  Determine novel genetic variants that indicate higher risk of disease progression and are associated with higher DTA scores.
Determine if DTA or any constituent radiomic features correlate with select plasma proteins. | 12 months
  MMP-7, CA-125, YKL, OPN, CCL18 are plasma proteins that have been shown to be associated with risk and prognosis in IPF.
Determine if DTA or any of constituent radiomic features correlate with transcriptomic | 12 months
  We have previously published a transcriptomic classifier that is predictive of FVC decline in IPF.
Determine the best combination of markers (DTA, proteins and transcriptome) for machine learning algorithms for AUC evaluation of ROCs on all 3 cohorts. | 12 months
  12-month FVC decline is a validated marker of disease progression in IPF as it's predictive of worse mortality. Receiver operating characteristic curve (ROC) is an analytical method, represented as a graph, that is used to evaluate the performance of a binary diagnostic classification method. The diagnostic test results need to be classified into one of the clearly defined dichotomous categories, such as the presence or absence of a disease. Area under the ROC curve (AUC) measures the entire two-dimensional area underneath the entire ROC curve.

SECONDARY OUTCOMES:
Determine associations of changes in DTA scores with 12-month changes in FVC and DLCO. | 12 months
  FVC (L) and diffusing capacity of the lungs for carbon monoxide (DLCO) have been shown to be validated markers of disease progression in IPF. DLCO is a measurement to assess the lungs' ability to transfer gas from inspired air to the bloodstream. The normal range for DLCO: 80-120% of its predicted value for men. 76-120% of its predicted value for women.
Determine associations of changes in DTA scores with drug treatment (i.e., antifibrotics) | 12 months
  Changes in DTA scores have been shown correlate strongly with changes in lung function. By establishing that changes in DTA scores occur in response to patients with IPF who start antifibrotic therapy, will provide supportive evidence of DTA as a potential tool to track treatment responses.

CONTACTS AND LOCATIONS:
Overall Officials: Noth Imre, MD, Principal Investigator — Division of Pulmonary and Critical Care; John Kim, Principal Investigator — Division of Pulmonary and Critical Care
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Plan to share de-identified dicom images with Ambrahealth for CT analysis

REFERENCES:
- [Background] Lederer DJ, Martinez FJ. Idiopathic Pulmonary Fibrosis. N Engl J Med. 2018 May 10;378(19):1811-1823. doi: 10.1056/NEJMra1705751. No abstract available. PMID 29742380
- [Background] Ley B, Ryerson CJ, Vittinghoff E, Ryu JH, Tomassetti S, Lee JS, Poletti V, Buccioli M, Elicker BM, Jones KD, King TE Jr, Collard HR. A multidimensional index and staging system for idiopathic pulmonary fibrosis. Ann Intern Med. 2012 May 15;156(10):684-91. doi: 10.7326/0003-4819-156-10-201205150-00004. PMID 22586007
- [Background] Podolanczuk AJ, Kim JS, Cooper CB, Lasky JA, Murray S, Oldham JM, Raghu G, Flaherty KR, Spino C, Noth I, Martinez FJ; PRECISIONS Study Team. Design and rationale for the prospective treatment efficacy in IPF using genotype for NAC selection (PRECISIONS) clinical trial. BMC Pulm Med. 2022 Dec 13;22(1):475. doi: 10.1186/s12890-022-02281-8. PMID 36514019
- [Background] Humphries SM, Swigris JJ, Brown KK, Strand M, Gong Q, Sundy JS, Raghu G, Schwarz MI, Flaherty KR, Sood R, O'Riordan TG, Lynch DA. Quantitative high-resolution computed tomography fibrosis score: performance characteristics in idiopathic pulmonary fibrosis. Eur Respir J. 2018 Sep 17;52(3):1801384. doi: 10.1183/13993003.01384-2018. Print 2018 Sep. PMID 30139770
- [Background] Humphries SM, Yagihashi K, Huckleberry J, Rho BH, Schroeder JD, Strand M, Schwarz MI, Flaherty KR, Kazerooni EA, van Beek EJR, Lynch DA. Idiopathic Pulmonary Fibrosis: Data-driven Textural Analysis of Extent of Fibrosis at Baseline and 15-Month Follow-up. Radiology. 2017 Oct;285(1):270-278. doi: 10.1148/radiol.2017161177. Epub 2017 May 10. PMID 28493789
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, Cottin V, Flaherty KR, Hansell DM, Inoue Y, Kim DS, Kolb M, Nicholson AG, Noble PW, Selman M, Taniguchi H, Brun M, Le Maulf F, Girard M, Stowasser S, Schlenker-Herceg R, Disse B, Collard HR; INPULSIS Trial Investigators. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2071-82. doi: 10.1056/NEJMoa1402584. Epub 2014 May 18. PMID 24836310
- [Background] Reichmann WM, Yu YF, Macaulay D, Wu EQ, Nathan SD. Change in forced vital capacity and associated subsequent outcomes in patients with newly diagnosed idiopathic pulmonary fibrosis. BMC Pulm Med. 2015 Dec 29;15:167. doi: 10.1186/s12890-015-0161-5. PMID 26714746
- [Background] Schmidt SL, Tayob N, Han MK, Zappala C, Kervitsky D, Murray S, Wells AU, Brown KK, Martinez FJ, Flaherty KR. Predicting pulmonary fibrosis disease course from past trends in pulmonary function. Chest. 2014 Mar 1;145(3):579-585. doi: 10.1378/chest.13-0844. PMID 24231810
- [Background] Paterniti MO, Bi Y, Rekic D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute Exacerbation and Decline in Forced Vital Capacity Are Associated with Increased Mortality in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2017 Sep;14(9):1395-1402. doi: 10.1513/AnnalsATS.201606-458OC. PMID 28388260